CLINICAL TRIAL: NCT03806569
Title: Mindfulness-Based Behavioural Group Therapy for Adult Attention Deficit Hyperactivity Disorder - Randomized Clinical Trial
Brief Title: MAC-cbt Group Therapy for Adults With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Tonn (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Peter Tonn, Director of the Center, Neuropsychiatrischen Zentrums Hamburg-Altona
Organization: Neuropsychiatrischen Zentrums Hamburg-Altona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUCHLER_2018
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Psychotherapy
Keywords: cognitive behavioral therapy; mindfulness; acceptance; commitment; adult ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: monocentric, parallel group randomized superiority study - one arm with new intervention, other arm with well established relaxation treatment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants will not know, in which of the arms they are; the outcomes assessor did not know the patients study-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAC-cbt group treatment for adult ADHD (Active Comparator): The patients will be treated with psychological group treatment for 8 sessions with focus on mindfulness, acceptance and commitment in a special adapted treatment process. This will be called "Mindfulness, Acceptance and Commitment-Therapy for adult Patients with ADHD"
  Interventions: Behavioral: MAC-cbt group treatment for adult ADHD
- Relaxation-group for adult ADHD (Sham Comparator): The patients will be treated with a relaxation-treatment, long-time established as "Jacobson muscle relaxing technique".
  Interventions: Behavioral: Jacobson

INTERVENTIONS:
Behavioral: MAC-cbt group treatment for adult ADHD — Psychotherapeutic intervention to treat adult patients with ADHD to be mindful, accept the symptoms and disturbances and commit with the situation or the possibility to change.
  Arms: MAC-cbt group treatment for adult ADHD
Behavioral: Jacobson — Relaxation treatment in technique of Jacobson in 8 sessions
  Arms: Relaxation-group for adult ADHD

SUMMARY:
The study is developed to validate a new short psychotherapeutic group treatment for adults with ADHD diagnosis. The participants will be treated in a monocentric, parallel group randomized superiority study - one group with the new treatment and one group with well established relaxing treatment.

DETAILED DESCRIPTION:
Background: Attention deficit hyperactivity disorder (AD(H)D) symptoms are often assumed to decease in adolescence, however in up to 60% of children, AD(H)D persists into adulthood. Currently, pharmacological therapy is the number-one choice AD(H)D treatment. Despite its evidenced effects of pharmacological interventions there are side effects, contraindications and non-responders, which send some patients disliking the use of medication and asking for alternative treatments. In previous studies mindfulness-based interventions already have shown similar effects in neural regions as pharmacological treatment and positive changes in AD(H)D symptoms, quality of life, awareness and concentration. The following study wants to improve mindfulness-based treatment approaches in AD(H)D with a new therapy concept.

Methods: Mindfulness, acceptance, commitment and cognitive behavioral group therapy (MAC-CBT) combines 3rd wave therapies with focus on mindfulness meditation, acceptance of unchangeability, commitment to new goals with elements of cognitive behavioral therapy. The design of this study is a single-center, parallel-group, randomized superiority trial. The aim is to compare MAC-CBT group with progressive muscle relaxation training (PMR by Jacobson). Both groups will be held over a period of eight weeks. Participants will be assessed two times before treatment to determine natural course of adult AD(H)D and two times after treatment to evaluate short and long term effects. A questionnaire battery and neuropsychological tests are to be used to obtain results regarding a possible change in the symptoms and attention, including selective attention.

Discussion: This trial will offer new knowledge about the effects of third wave therapies on AD(H)D. Furthermore, the following study is one of few studies that will compare AD(H)D treatment to relaxation training instead of comparison to waiting list. The aim of the following study is to verify previous outcomes of mindfulness-based treatments on AD(H)D and to evaluate superiority of mindfulness towards relaxation programs.

ELIGIBILITY:
Inclusion Criteria:

* adult ADHD
* written informed consent
* stable medication for at least two weeks
* sufficient knowledge of the German language

Exclusion Criteria:

* personality disorder
* schizophrenia / psychotic disorders
* bipolar disorder
* acute suicidality
* disease of the central nervous system
* no other psychotherapeutic treatment at the time of the study
* pregnancy
* IQ below 70 Points

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change of Symptoms measured by the Connors ADHD Adult Rating Scale (CAARS) | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  The long version of the CAARS (Conner's Adult AD(H)D Rating Scales (Christiansen et al., 2012)) combines self-report and observer rating questionnaires to assess current AD(H)D symptoms in adulthood. This instrument consists of 66 items based on a 4-point Likert scale and four subscales: Inattention/ Memory Problems, Hyperactivity/ Restlessness, Impulsivity/ Emotional Lability and Problems with Self-Concept. With regard to the scientific quality criteria, Christiansen (2012) reports internal consistencies with a Cronbach's α of .74 to .95 and a test-retest reliability from .71 to .93, range min. 66 to max. 264 points.

SECONDARY OUTCOMES:
Measure of the quality of life of the participants measured by World Health Organization Quality of Life Questionnaire | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  Quality of life will be assessed by the short version of WHOQOL-BREF (World Health Organization Quality of Life Questionnaire (Group, 1998)). The questionnaire consists of 26 items that were extracted from the complete version consists of 100 items (WHOQOL-100) based on a 5-point Likert scale. For the German short version, Cronbach's alpha scores between .76 and .88 (Skevington, Lotfy, O'Connell, & Group, 2004). Range from 26 to 105 (min.-max).
Changes of attention functioning measured by change detection task and trail making test A and B of the computer based test setting Psychology Experiment Building Language (PEBL) | Measurement 1 at inclusion , Measurement 2 is 2 months after inclusion, measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  The change detection task, modeled paradigm by Luck and Vogel, examines the visual working memory and covers sustained and selective attention. Patients will see a first pattern of differently colored squares for 300ms followed by a 1000ms pause and then a second pattern of squares. The task is then to determine whether the colors of every square are identical, will be repeated 120 times and takes approximately 12 minutes in total. Reaction times and the amount of mistakes made will then give information on the level of functioning. In addition, a TMT-A and B (Reitan, 1992) will be conducted. Patients will be asked to first connect numbers ranging from 1 to 30 in increasing order and then numbers from one to 15 and letters from A through O alphabetically alternating. Reaction times, times between clicks and the amount of correct and incorrect clicks will provide insight to the level of attentional functioning. Measurement of single individual scores, no qualified range described.
Changes of mindfulness measured by Mindful Attention Awareness Scale | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  In order to assess mindfulness as well as the perception of the "here and now", the German version of the MAAS (Mindful Attention Awareness Scale (Brown & Ryan, 2003)) is used. In total, it consists of 15 items on a 6-point Likert scale. Since non-mindful behaviors are described, high scores mean a higher level of mindfulness. The internal consistency, represented by Cronbach's alpha, amounts α = .83 for the German version (Michalak, Heidenreich, Ströhle, & Nachtigall, 2008).Range form 15 to 90 points.
Changes of acceptance, measured by Acceptance and Action Questionnaire | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  The FAH II Questionnaire (Acceptance and Action Questionnaire), the German version of AAQ (Acceptance and Action Questionnaire (Bond et al., 2011; Hoyer & Gloster, 2013)), aims to measure acceptance and psychological flexibility. The questionnaire consists of seven items, based on a 7-point Likert scale. Hoyer and Gloster found Cronbach's alpha between.84 and .97 and a test-retest reliability of rtt = .74 - .85 for the German version (2011). Range from 7 to 49 points.
Affective state measured with the Patient Health Questionnaire PHQ-9 | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  The PHQ (Patient Health Questionnaire, (Gräfe, Zipfel, Herzog, & Löwe, 2004)) is used for psychodiagnostic screening and a possible change in patient depression. It is a self-assessment tool based on the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV (Saß & Association, 1998)) and includes modules on somatoform disorders, depressive disorders, anxiety disorders, and eating disorders, alcohol abuse, psychosocial functioning, stressors, critical life events and for participants to menstruation, pregnancy and childbirth. In total, it contains 78 items, which are based on a 2- to 5-point Likert scale depending on the module. For the depression scale of PHQ-D the internal consistency according to Cronbach's alpha is α = .88, for the somatization scale α = .79. Different subscales, no combined score, individual ranges and scores.
Measuring of satisfaction and willingness to change with visual analogue scales | Measurement 1 at inclusion date, Measurement 2 two months later measurement 1, then measurement 3 immediately after intervention, measurement 4 as catamnestic follow up 6 months after intervention
  Visual analogue scales (VAS) with regard to satisfaction with mental health and the willingness to change are going to be evaluated.Range from 0 to 10 per scale, no combined scores.
Measuring of five individual parameters during every of the single treatment session | Measurement before and after every treatment session, 2-6 weeks after inclusion date, every week for the 8 weeks treatment period
  Each time before and after the therapy sessions, five visual analogue scales are to be filled in, on which patients evaluate their current mood, stress, restlessness, trust in effectiveness of psychotherapy and their energy level. Range from 0 to 10 per scale, no combined scores.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Moritz, Prof., Principal Investigator — UKE Hamburg; Peter Tonn, Dr. med., Principal Investigator — NPZ Hamburg
Locations (1):
- Neuropsychiatric Center of Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No